CLINICAL TRIAL: NCT03561948
Title: Feasibility of Intraperitoneal Chemotherapy in the Surgical Treatment of Colon Cancer cT4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State Scientific Centre of Coloproctology, Russian Federation (Other Government)
Responsible Party: Principal Investigator, Achkasov Sergey, Professor Sc.State Scientific Centre of Coloproctology, Head of Surgical department of sugery and oncology of colon, Moscow,Russian Federation, State Scientific Centre of Coloproctology, Russian Federation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13
Record Dates: First submitted 2018-05-30; First posted 2018-06-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Colon Cancer
Keywords: intraperitoneal chemotherapy; Peritoneal Carcinomatosis; Colonic Diseases
MeSH Terms: conditions — Colonic Neoplasms; Peritoneal Neoplasms; Colonic Diseases | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Surgery and Intraperitoneal Chemotherapy
  Interventions: Procedure: Experimental group
- Control group (Placebo Comparator): only surgery
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: Experimental group — After performing the surgical intervention, the patient will undergo intraoperative intra-abdominal chemotherapy with mitomycin C. Further, lavage of the abdominal cavity will be repeated, followed by immunological examination.
  Arms: Experimental group
Procedure: Control group — In the control group (40 patients), after laparotomy and revision, peritoneal lavage will also be performed with subsequent immunological examination. Patients of this group will not receive intraperitoneal chemotherapy. After performing the surgical intervention, the patient will be irrigation of the abdominal cavity with physiological saline. Further, lavage of the abdominal cavity will be repeated, followed by immunological examination.
  Arms: Control group

SUMMARY:
This is a randomised controlled study aims to determine the oncological effectiveness of adjuvant HIPEC, using intraperitoneal Mytomicin C following a curative resection of a cT4 Colon cancer in preventing the development of peritoneal carcinomatosis in addition to the standard adjuvant systemic treatment.

DETAILED DESCRIPTION:
In the experimental group (50 patients) after laparotomy and revision of the abdominal cavity organs, peritoneal lavage will be performed followed by immunological examination. After performing the surgical intervention, the patient will undergo intraoperative intra-abdominal chemotherapy with mitomycin C. Further, lavage of the abdominal cavity will be repeated, followed by immunological examination.

In the control group (40 patients), after laparotomy and revision, peritoneal lavage will also be performed, followed by immunological examination. Patients of this group will not receive intraoperative intra-abdominal chemotherapy. After performing the surgical intervention, the patient will perform irrigation of the abdominal cavity with physiological saline. Further, lavage of the abdominal cavity will be repeated, followed by immunological examination.

ELIGIBILITY:
Inclusion Criteria:

1. Colon cancer which represent cT4N0-2 M0 on the basis of preoperative examination data (CT of the chest, abdominal and pelvic organs) in line with The American Joint Committee on Cancer: the 7th edition of the AJCC cancer staging manual:
2. Histologically verified adenocarcinoma of the colon.
3. Signed informed consent.

Exclusion Criteria:

1. Pregnancy or lactation.
2. The presence of synchronous or metachronous malignant tumors.
3. Distant metastases to the liver, lungs, peritoneal carcinomatosis and other organs.
4. Neoadjuvant chemotherapy.
5. Suspected Lynch syndrome.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
Positive peritoneal lavage | through study completion, an average of 1 year
  Cancer cell vitality

CONTACTS AND LOCATIONS:
Locations (1):
- State Scientific Centre of Coloproctology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No